CLINICAL TRIAL: NCT03672357
Title: Short and Long Outcomes Between Laparoscopic and Open Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hui hou (Other)
Responsible Party: Sponsor-Investigator, hui hou, Director of the hepatobiliary surgery department, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LLR_01
Record Dates: First submitted 2018-08-19; First posted 2018-09-14 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Laparoscopic Liver Resection; Open Liver Resection
Keywords: Liver resection; Laparoscopic surgery; fast recovery

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic liver resection (Experimental): Laparoscopic hepatectomy
  Interventions: Procedure: Laparoscopic liver resection
- Open liver resection (Other): Open hepatectomy
  Interventions: Procedure: Open liver resection

INTERVENTIONS:
Procedure: Laparoscopic liver resection — Laparoscopic hepatectomy
  Arms: Laparoscopic liver resection
Procedure: Open liver resection — Traditional open hepatectomy
  Arms: Open liver resection

SUMMARY:
LLR was applied for tumors located at the lower edge and lateral segments of the liver that could be resected more easily than posterosuperior segments. With the development of technology and the growing experience of hepatobiliary surgeons, LLR has been expanded to major liver resections, anatomical resections, and donor hepatectomies by skilled surgeons. However, due to the concerns over the risk of operative bleeding, tumor seeding and positive resection margin, the true benefit of LLR remains unclear across surgical community.

DETAILED DESCRIPTION:
The 2nd International Consensus Conference on Laparoscopic Liver Resection (ICCLLR) was held in Morioka, Japan, in 2014. The new recommendations of the ICCLLR state that the outcomes of LLR are not inferior than OLR regarding to operative mortality rate and margin negativity, and are superior in decreasing postoperative complications, blood loss, and the length of the postoperative hospital stay. However, it is not clear that whether LLR is able to alleviate the impairment of liver function after hepatic resection, and there is no RCTs to compare the short and long outcomes between LLR and OLR.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who underwent hepatectomy for benign or malignant neoplasm of the liver, and is suitable for both open and laparoscopic liver resection;
2. Child-Pugh A without portal hypertension
3. No portosystemic shunt
4. No previous abdominal operation history.
5. American society of anesthesiology class(ASA): I or II
6. Age 18 to 80

Exclusion Criteria:

1. Additional intervention to the liver (Radio Frequent Ablation, Percutaneous Ethanol. Injection Therapy or others)
2. Combined hepatectomy
3. Intrahepatic duct stone disease
4. Liver disease caused splenomegaly
5. Previous hepatectomy
6. Combined operation for extrahepatic disease
7. Vulnerable population (mental retardation, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of serum glutamic oxalacetic transaminase | up to 7 days after liver resection
  Change of serum glutamic oxalacetic transaminase after liver resection.These values will be recorded preoperative, and postoperative day-1,3,5,7.
Change of serum glutamic-pyruvic transaminase | up to 7 days after liver resection
  Change of serum glutamic-pyruvic transaminase after liver resection.These values will be recorded preoperative, and postoperative day-1,3,5,7.

SECONDARY OUTCOMES:
Postoperative complication(Rates in different grades) | up to 30 days after liver resection
  According to The Clavien-Dindo Classification, https://www.assessurgery.com/clavien-dindo-classification/
Mortality rates | up to 30 days after liver resection
  the rate of postoperative death
Hospital duration after operation (days) | up to 30 days after liver resection
  the length of hospital stay
Operation time(min) | up to 30 days after liver resection
  the during of operation
Blood loss(ml) | up to 30 days after liver resection
  the volume of blood loss
Blood transfusion (times and units) | intraoperative
  intraoperative blood transfusion
Duration of nasogastric tubes (hours) | up to 14 days after liver resection7
  Duration of nasogastric tubes
Duration of abdominal drain (days) | up to 14 days after liver resection
  Duration of abdominal drain
Duration to first flatus (days) | up to 14 days after liver resection
  Duration to first flatus
Comfort questionnaire measures (GCQ) measures by Kolcaba | up to 7 days after liver resection
  GCQ measures by Kolcaba, download from http://www.thecomfortline.com/resources/cq.html.
Resection margin status | up to 30 days after liver resection
  the R0 resection rate
Intensive care unit stay (days) | up to 7 days after liver resection
  Intensive care unit stay in days
Readmission rate | up to 30 days after liver resection
  measure the rate of readmission
C-reactive protein (mg/mL) | up to 5 days after liver resection
  C-reactive protein levels on preoperative and postoperative day-1,3,5
Disease recurrence rates | up to 5 years
  The disease recurrence after operation
Overall survival time (month) | up to 5 years after operation
  Overall survival time after operation
Disease free survival time (month) | up to 5 years after operation
  Disease free survival time after operation

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Anhui Medical University,, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No